CLINICAL TRIAL: NCT00260325
Title: Effect of Valdecoxib Pretreatment on Pain and Secondary Hyperalgesia: a Randomized Controlled Trial in Healthy Volunteers
Brief Title: Effect of Valdecoxib Pretreatment on Pain and Secondary Hyperalgesia in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Pfizer (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 70,328-01; IIG Pfizer(PJK); MOIRR10732
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Pain; Hyperalgesia
Keywords: pretreatment; healthy volunteers
MeSH Terms: conditions — Pain; Hyperalgesia | interventions — valdecoxib

INTERVENTIONS:
Drug: valdecoxib

SUMMARY:
Tis study was designed to test the hypothesis that pretreatment with valdecoxib, prior to injury could reduce or prevent the development of secondary hyperalgesia around the area of primary injury. A heat/capsaicin model of induced hyperalgesia was tested in healthy volunteers in a randomized, double blind, cross-over trial of a single dose of 40 mg vadecoxib versus control. Subjects rated pain intesnsity and unpleasantness following heat stimulation of the forearm, the area of hyperalgesia was also mapped over the course of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* healthy male of non-pregnant female; 18yo or older
* not currently taking NSAID
* able and willing to provide informed consent
* willing to avoid other NSAIDs in 24 hour period following study
* no known hypersentitivites or contraindications to NSAIDS, sulfonomides or capsaicin

Exclusion Criteria:

* pregnant or breast feeding
* use of NSAIDS or other analgesic medications in past 7 days
* unwilling or unable to give informed consent
* contraindication to any study medication or other NSAID

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-08; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Reduction in the area of secondary hyperalgesia

SECONDARY OUTCOMES:
Reduction in pain threshold
Reduction in pain unpleasantness

CONTACTS AND LOCATIONS:
Overall Officials: Piotr K Janicki, MD, PhD, Principal Investigator — Penn State University, Dept of Anesthesiology
Locations (1):
- Penn State University College of Medicine, Hershey, Pennsylvania, United States